CLINICAL TRIAL: NCT04233684
Title: Rapid Urease Test for Helicobacter Pylori in Population Who Stop Proton Pump Inhibitor Less Than 2 Weeks Compared With Histology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principle investigator, King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP015
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Masking Description: The pathologists will be blinded for the result of endoscopic finding and rapid urease test.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study (Experimental): * Rapid urease test is the test for H. pylori infection by detect the change of pH by urease enzyme metabolism.
  * Pathologic test for H. pylori by H&E stain and Giemsa stain
  * All tissues will be sent to immunohistochemistry as a gold standard
  Interventions: Diagnostic Test: rapid urease test

INTERVENTIONS:
Diagnostic Test: rapid urease test — Rapid urease test is the test for H. pylori infection by detect the change of pH by urease enzyme metabolism.
  Pathologic test for H. pylori by H&E stain and Giemsa stain Gold standard is a immunohistochemistry.
  Other Names: pathologic test

SUMMARY:
Patients with dyspepsia will have negative impact to their life and common cause is Helicobactor pylori infection. Rapid urease test is the easy available and rapid method to test the infection but the test may be interfered by proton pump inhibitor, bismuth or antibiotics .In general, patients with dyspepsia usually take proton pump inhibitor to relieve dyspepsia so those patients may not stop the drug before test the infection with rapid urease test. So author aims to measure the sensitivity of rapid urease test from biopsy of body, which H. pylori would migrate if the patients still take proton pump inhibitor and biopsy of antrum, which is standard location of biopsy compare to pathology for H. pylori in each sites in patients who do not stop taking proton pump inhibitor

DETAILED DESCRIPTION:
The investigators contacted patients who had an appointment for esophagoendoscopy(EGD) at Chulalongkorn Hospital to inform and review patient's history. If patients matched inclusion and did not meet exclusion criteria, the participants would tell the information of the study including proposal, method, risk and benefit then the investigators asked for consent to participate in the study.

If patients decided to participate then the investigator corrected the information in CRF form which was sex, age, underlying disease, smoking history, alcohol drinking history, current and past medication especially PPI and NSIADs, EGD and rapid urease test history, H. pylori treatment history, duration of taking PPI drug.

EGD was done by endoscopist with standard method. The investigator performed biopsy at antrum, 5 cm proximal to pylorus lesser curvature, and body, greater curvature opposite to angularis by standard forceps. The biopsy would take 2 times from each site for rapid urease test and histopathology test for H. pylori. The endoscopists change forceps after finishing biopsy in each site to reduce contamination. The EGD finding was recorded After the investigators test H. pylori by rapid urease test, the result was read at 24 hours at room temperature. The color changing from yellow to pink was positive test, which mean there was H. pylori infection. In contrast, negative test was no color changing.

For Histopathologic test, the investigators fixed sample in formalin, infiltrated the tissue with paraffin then embedded. Stained with Hematoxylin & Eosin and looked for H. pylori by 2 histopathologists, who were blinded the result to each other and result of rapid urease test. If negative study, the histopathologists would stain tissue with giemsa and corrected data again. All gastric tissue will be sent for immunohistochemistry as a gold standard for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspepsia and have indication for esophagogastroscopy
* Patients who take PPI at least 2 weeks and stop the drug less than 2 weeks
* Age above 18 years old

Exclusion Criteria:

* Patients who diagnosed to have iron deficiency anemia and have signs of previously bleeding gastric ulcer
* Active upper gastrointestinal bleeding or recent bleeding
* previous gastric surgery
* patients who take bismuth or antibiotic in last 4 weeks
* Coagulopathy, INR>1.5, Platelet < 100,000
* gastric cancer
* Life expectancy less than 3 months
* Deny to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of rapid urease test for dectection of H.pylori from gastric antrum and body | 24 hours after test by rapid urease test
  The sensitivity of rapid urease test for H.pylori diagnosis at antrum, body and both in patients stopping proton pump inhibitors less than 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pittayanon Pittayanon, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, State/Region/Province/District, Thailand